CLINICAL TRIAL: NCT04565379
Title: A Randomized, Double Blind, Placebo-controlled, Phase 2 Clinical Trial to Investigate the Efficacy and Safety of 2 Doses of NuSepin® Intravenous Infusion in COVID-19 Pneumonia Patients
Brief Title: Clinical Trial to Investigate the Efficacy and Safety of NuSepin® in COVID-19 Pneumonia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaperon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shaperon001; 2020-003107-34 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID19 Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NuSepin® 0.1 mg (Active Comparator): NuSepin® 0.1 mg/kg in 100 ml normal saline infusion
  Interventions: Drug: NuSepin® 0.1 mg
- NuSepin® 0.2 mg (Active Comparator): NuSepin® 0.2 mg/kg in 100 ml normal saline infusion
  Interventions: Drug: NuSepin® 0.2 mg
- Placebo (Placebo Comparator): 100 ml normal saline infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NuSepin® 0.1 mg — NuSepin® 0.1 mg
  Arms: NuSepin® 0.1 mg
Drug: NuSepin® 0.2 mg — NuSepin® 0.2 mg
  Arms: NuSepin® 0.2 mg
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
A randomized, double blind, placebo-controlled, phase 2 clinical trial to investigate the efficacy and safety of 2 doses of NuSepin® intravenous infusion in COVID-19 pneumonia patients

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects aged between 18≤ and <80 years old
2. Laboratory-confirmed SARS-CoV-2 infection by PCR test for the first time within 144 hours prior to randomization
3. Diagnosis of pneumonia based on:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan) AND
   * 3 of the following clinical symptoms: new onset cough, fever, fatigue, sputum (all day), tachypnea, dyspnea, pleuritic chest pain AND
   * CRP value > 10 mg/L
4. Patients with blood leukocyte count > 4.0 x 109 /L and lymphocyte count > 0.7 x 109

   * L
5. Patients with SpO2 ≤ 94% on room air or Pa02/FI02 ratio < 300mgHg at screening
6. Patients capable to give consent and who have signed the informed consent form before any trial related assessment.
7. Medically accepted effective contraception for women of childbearing potential (WOCBP) which should be continued until at least 90 days after the last dose of trial treatment.
8. Patients with NEWS2 score > 7

Exclusion Criteria

1. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
2. Reduced renal function with estimated glomerular filtration rate (eGFR) < 30 ml/min or hemodialysis or hemofiltration.
3. Pregnancy or breast feeding.
4. Evidence of multiorgan failure
5. Steroid treatment by any reason within 72 hours prior to enrolment
6. Participation in any other clinical trial of an experimental agent treatment for COVID-19
7. Physician makes a decision that trial involvement is not in patients' best interest, or any condition that does not allow the protocol to be followed safely.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Difference in Time to Clinical Improvement (TTCI) between the 2 treatments and the placebo group (in days) | Day 29

SECONDARY OUTCOMES:
Percentage of patients with CRP < 10 mg/L or < 30% decreases from baseline | Day 15 and Day 29
Clinical Status assessed by the six-category ordinal scale at fixed time points | Day 1, 4, 9, 15 and 29
  Minimum value being 1, Maximum value being 6. Smaller the number, better the clinical status & outcome
Time to complete clinical remission OR NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hours | Up to Day 29
All-cause mortality | Up to Day 29
Duration (days) of mechanical ventilation | Up to Day 29
Duration (days) of extracorporeal membrane oxygenation | Up to Day 29
Duration (days) of supplemental oxygenation | Up to Day 29
Length of hospital stay (days) | Up to Day 29
Length of ICU stay (days) | Up to Day 29
Number of incidence of treatment emergent adverse events (TEAEs) in 3 treatment groups | Day 15 and Day 29

OTHER OUTCOMES:
Serum level of TNF-α in pg/ml | Day 0, 4, 9, 15 and 29
Serum level of IL-1β in pg/ml | Day 0, 4, 9, 15 and 29
Serum level of IL-6 in pg/ml | Day 0, 4, 9, 15 and 29
Serum level of IL-8 in pg/ml | Day 0, 4, 9, 15 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yong Seong, Dr., Study Chair — Shaperon Inc.
Locations (5):
- Romania (5):
  - "Leon Daniello" Clinical Hospital of Pneumophtisiology Cluj-Napoca Pneumology Clinic, Cluj-Napoca
  - Clinical Hospital for Infectious Diseases and Pneumophtisiology "Victor Babes", Craiova Infectious Diseases Clinic for Adults, Craiova
  - "Sf. Parascheva" Infectious Diseases Clinical Hospital Iasi Infectious Diseases Department, Iași
  - Ramnicu Sarat Clinical Hospital, Râmnicu Sărat
  - "Sf. Ioan cel Nou" Suceava County Emergency Hospital Infectious Diseases Department, Suceava